CLINICAL TRIAL: NCT00852215
Title: Do Cobalt Chrome Stent and Paclitaxel-Eluting Stent Have Equivalent Clinical Result in Non-Complex Lesion? (COPE Study): Long-Term Follow-up Study
Brief Title: Do Cobalt Chrome Stent and Paclitaxel-Eluting Stent Have Equivalent Clinical Result in Non-Complex Lesion?
Acronym: COPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: HC Gwon, MD, PhD / Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-07-014
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; Paclitaxel-eluting stent; Vision stent
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- 1 (Active Comparator): Taxus stent group
  Interventions: Device: Taxus stent
- 2 (Active Comparator): Vision stent group
  Interventions: Device: Vision stent

INTERVENTIONS:
Device: Taxus stent — Stenting with Paclitaxel-eluting coronary stent system for coronary lesions with > 50% diameter stenosis with ischemic symptoms or positive functional study, or > 70% diameter stenosis without ischemic symptoms or positive functional study
  Arms: 1
Device: Vision stent — Stenting with VISION coronary stent system for coronary lesions with > 50% diameter stenosis with ischemic symptoms or positive functional study, or > 70% diameter stenosis without ischemic symptoms or positive functional study
  Arms: 2

SUMMARY:
We sought to evaluate the long-term safety and efficacy of drug-eluting stent in large vessels compared with bare metal stent.

DETAILED DESCRIPTION:
Drug-eluting stent (DES) has been proved to reduced restenosis rate dramatically compared to bare metal stent (BMS). However, the long-term safety of DES is still uncertain. Recent meta-analysis showed that very late stent thrombosis rate was higher in DES group although overall mortality was similar between 2 groups.

The safety issue of DES was first suggested in the BASKET-LATE study, which compared cobalt chromium alloy BMS (VISION®, Guidant, USA) with sirolimus- or paclitaxel-coated DES. The study showed a significantly higher rate of death or myocardial infarction in the DES group between 7 and 18 month after the procedure (BMS 1.3%, DES 4.9%, p=0.01). Moreover, benefit to reduce target vessel revascularization was not found and there was even the possibility of late harm in patients treated with DES in large native vessels.

We perform a multicenter prospective randomized study comparing paclitaxel-eluting stent with cobalt chromium stent several years, originally to see whether major adverse cardiac event is significantly lower in DES compared to thin-strut BMS in the non-complex lesion subset. In this article, we would like to investigate the 2-year clinical events in DES and BMS groups.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically proved significant stenosis in native coronary artery (> 50% diameter stenosis with ischemic symptoms or positive functional study, or > 70% diameter stenosis without ischemic symptoms or positive functional study)
* planned target lesion number =< 2
* reference diameter 2.75 - 4.0 mm
* lesions can be fully covered by one 28 mm or shorter stent

Exclusion Criteria:

* unprotected left main coronary disease with more than 50% stenosis or planned left main angioplasty
* ostial target lesion (within 5 mm of ostium)
* angiographic evidence of thrombus within target lesion
* calcified lesions which cannot be successfully predilated
* instent restenosis
* multi-vessel intervention more than 2 lesions
* atherectomy is planned before stenting
* bifurcation lesion that needs side branch ballooning or stenting
* Severe left ventricular dysfunction with echocardiographic ejection fraction less than 30%
* ST-elevation myocardial infarction within the preceding 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE: cardiac death, myocardial infarction, or target vessel revascularization) | 1 year

SECONDARY OUTCOMES:
MACE and stent thrombosis by the criteria of Academic Research Consortium | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea